CLINICAL TRIAL: NCT05745285
Title: The Impact of a Non-Profit Cancer Advocacy Organization on Patient Reported Outcomes and Access to Care: A Multisite, Longitudinal Trial
Brief Title: Leukemia and Lymphoma Society (LLS) Services Impact on Outcomes and Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Frank Penedo, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20220784; 20220220 (Other: University of Miami)
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Leukemia; Lymphoma; Myeloma; Myelodysplastic Syndromes; Myeloproliferative Neoplasm
Keywords: Blood cancer
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myeloproliferative Disorders; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLS Program and Usual Care Group (Experimental): Participants in the LLS Program and Usual Care condition will receive LLS services such as information, services, and financial aid so that patients can have better access to healthcare and better quality of life. Participants will also receive the standard care. Participants will be in this group for 6 months.
  Interventions: Other: LLS Program
- Usual Care Group (No Intervention): Participants will receive the standard care. Participants will be in this group for 6 months.

INTERVENTIONS:
Other: LLS Program — The intervention will be conducted virtually. Participants will receive LLS's free patient and caregiver services including co-pay assistance, transportation and urgent need assistance, a scholarship program for young adult patients and survivors, one-on-one peer-to-peer support, online chats and support groups facilitated by clinical social workers, and nutrition counseling with a registered dietician for 6 months.
  Arms: LLS Program and Usual Care Group

SUMMARY:
The purpose of this study is to learn about the impact that the services and programs provided by the Leukemia and Lymphoma Society have among patients with blood cancer, such as access to care, quality of life, and financial burden.

ELIGIBILITY:
Inclusion Criteria:

* Be currently receiving primary or relapse treatment for a diagnosis of leukemia, lymphoma, myeloma, myelodysplastic syndromes (MDS), or myeloproliferative neoplasms (MPN)
* Report experiencing at least one unmet need addressed by the LLS Program (i.e., medical care including second opinions, travel for care, clinical trial access, financial and insurance needs, supportive programs, disease and treatment education)
* Not be currently participating in any LLS programs or services
* Be willing to be followed for 6 months
* Speak English or Spanish

Exclusion Criteria:

* Are not receiving primary or relapse treatment for a diagnosis of leukemia, lymphoma, myeloma, myelodysplastic syndromes (MDS), or myeloproliferative neoplasms (MPN)
* Are not experiencing unmet needs addressed by the LLS Program (i.e., medical care including second opinions, travel for care, clinical trial access, financial and insurance needs, supportive programs, disease and treatment education)
* Are currently participating in any LLS programs or services
* Are not willing to be followed for 6 months
* Do not speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of care needs as measured by the Access to Care Survey | Baseline, 3 month, 6 month
  Change in number of care needs will be assessed via the self-report Access to Care Survey which includes access to primary and specialty care, access to medications specific to cancer care, and access to financial resources specific to cancer care. The survey uses a composite score to assess participants' needs. Scores range from 0 to 21 with lower scores indicating better access to care needs.
Change in number of medication access problems as measured by the Access to Care Survey | Baseline, 3 month, 6 month
  Change in number of medication use will be assessed via the self-report Access to Care Survey which includes access to medications specific to cancer care. The survey uses a composite score to assess participants' medication use. Scores range from 0 to 6 with lower scores indicating better access to medication.

SECONDARY OUTCOMES:
Change in general health-related quality of life (HRQL) | Baseline, 3 month, 6 month
  The Functional Assessment of Cancer Therapy-General (FACTG) 5 will be administered to evaluate general domains of HRQL. Quality of life is scored on a scale with scores ranging from 0 to 108, with higher scores indicating better health-related quality of life outcomes.
Change in treatment satisfaction as measured by FACIT | Baseline, 3 month, 6 month
  The 8-item Functional Assessment of Chronic Illness Therapy (FACIT) Treatment Satisfaction - General (TS-G) is a Likert scale designed to assess satisfaction with general medical treatments. A summary score yields a treatment satisfaction composite with higher scores indicating greater treatment satisfaction.
Change in financial toxicity as measured by FACIT-COST | Baseline, 3 month, 6 month
  The 12-item Functional Assessment of Chronic Illness Therapy - Comprehensive Score for Financial Toxicity (FACIT-COST) is a patient reported outcome measure that describes the financial distress experienced by cancer patients. Score range 0-44 with higher scores indicating better Financial Well-Being.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Penedo, PhD, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Mays Cancer Center at UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No